CLINICAL TRIAL: NCT01386671
Title: Safety and Efficacy of Metformin Glycinate vs Metformin Hydrochloride on Metabolic Control and Inflammatory Mediators in Type 2 Diabetes Patients
Brief Title: Metformin Glycinate on Metabolic Control and Inflammatory Mediators in Type 2 Diabetes
Acronym: COMET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GlyMet01_13062011
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; metformin glycinate; metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin glycinate (Experimental): Metformin glycinate is a new biguanide, for this study the dose administrated will be 1050.6 mg OD for a month, and 1050.6 mg BID for 11 moths.
  Interventions: Drug: Metformin glycinate
- Metformin Hydrochloride (Active Comparator): Metformin Hydrochloride is the biguanide most used, for this study the dose administrated will be 850 mg OD for a month, and 850 mg BID for 11 months.
  Interventions: Drug: Metformin hydrochloride

INTERVENTIONS:
Drug: Metformin glycinate — Drug: Metformin glycinate 12 months: 1 month,one tablet 1050.6 mg once daily + 11 months, one tablet 1050.6 mg twice daily
  Arms: Metformin glycinate
Drug: Metformin hydrochloride — 12 months: 1 month, once daily dose of 850 mg (before dinner) and 11 months, twice daily dose 850 mg (before breakfast) + 850 mg (before dinner).
  Other Names: Predial
  Arms: Metformin Hydrochloride

SUMMARY:
The aim of this study is to compare the efficacy and safety of Metformin Glycinate versus Metformin Hydrochloride in metabolic control and inflammatory mediators in Mexican type 2 diabetes patients, in a 12 months follow up.

DETAILED DESCRIPTION:
Metformin glycinate salt is a new drug , which has better pharmacokinetic characteristics (better bioavailability and absorption) making a proper antihyperglycemic power without increasing the frequency of adverse effects. The drug has been tested in preclinical test with animals, in healthy subjects and in patients with type 2 diabetes; which showed that it has adequate antihyperglycemic effect. Now, its important to compare metformin glycinate and metformin hydrochloride for evaluate the relative antihyperglicemic power. In addition, a study with a larger number of patients improve the statistical power of the test to investigate the effects of these drugs on possible weight loss and lipid profile improve. Additionally, it will also explore the relative power of the two medications tested to modify inflammatory response mediators and oxidative stress have been associated with the incidence of cardiovascular disease in diabetes. This project was designed with the intent to answer the next question: What are the efficacy and safety of metformin glycinate dose of 2101.2 mg/day (equivalent to 1700 mg/day metformin hydrochloride), compared with metformin hydrochloride in doses of 1700 mg/day for 12 months of treatment in patients with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes according ADA
* Less than a year of evolution since diagnosis
* Without antihyperglycemic pharmacological treatment
* HbA1c between 6.5% and 9.5%
* Stable weight during the last 6 months
* Body Mass Index ≥ 25 kg/m2 and <35kg/m2.
* Blood pressure ≤ 130/80 mmHg
* Childbearing women under contraceptive treatment
* Signed Informed Consent Form
* Age from 18 to 70 years old

Exclusion Criteria:

* Non-fulfilment treatment in the screening period
* Smoking up to 1 year before the initial examination
* Drugs or alcohol abuse
* Creatinine depuration estimated with MDRD formula using serum creatinine < 90 ml/min/1.72m2
* History of chronic liver disease, ALT or AST ≥ 2 times from the normal superior limit, or GGT ≥ 3 times from the normal superior limit.
* Chronic lung disease, that causes dyspnea equivalent to a functional class ≥3 (NYHA)or that requires oxygen supplementation.
* History or symptoms of coronary artery disease (CAD) or cerebrovascular disease (CVD).
* Drug treatment that interact with biguanides.
* Another chronic diseases that restricts survival or associated with chronic inflammation like: cancer, leukemia, lymphoma, erythematosus lupus, asthma, rheumatoid arthritis or infection for HIV.
* Pregnancy or positive pregnancy test in women under 50 years old or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) | 12 months
  HbA1c: Measured by electrophoresis of lacked total blood using Paragon system and Appraise reader 44800 (Beckman Instruments de Mexico).
  Fasting Glucose: in serum using glucose oxidase technique with BM/Hitachi 704/911 automated analyzer

SECONDARY OUTCOMES:
Fasting glucose | 12 months
Total cholesterol | 12 months
High-density lipoprotein (HDL) | 12 months
Low-density lipoprotein (LDL) | 12 months
Triglycerides | 12 months
Tumor necrosis factor-alpha (TNF-α) | 12 months
Adiponectin | 12 months
Resistin | 12 months
Interleukin-1 beta (IL-1β) | 12 months
Number of Adverse Events as a Measure of Safety and Tolerability | 12 months
Malonylaldehyde | 12 months
Dismutase superoxide | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Niels H Wacher, PhD, Principal Investigator — IMSS
Locations (4):
- Mexico (4):
  - Paracelsus S.A. de C.V., Mexico City, AA
  - Unidad Antidiabética Integral, Mexico City, AA
  - Instituto de terapéutica experimental y clínica (INTEC), Guadalajara, Jalisco
  - Unidad de Investigacion en Epidemiologia Clinica. UMAE Hospital de Especialidades Centro Medico Nacional Siglo XXI. Instituto Mexicano del Seguro Social, Mexico City, Mexico City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hermann LS, Schersten B, Melander A. Antihyperglycaemic efficacy, response prediction and dose-response relations of treatment with metformin and sulphonylurea, alone and in primary combination. Diabet Med. 1994 Dec;11(10):953-60. doi: 10.1111/j.1464-5491.1994.tb00253.x. PMID 7895460
- [Background] Johnson JA, Simpson SH, Toth EL, Majumdar SR. Reduced cardiovascular morbidity and mortality associated with metformin use in subjects with Type 2 diabetes. Diabet Med. 2005 Apr;22(4):497-502. doi: 10.1111/j.1464-5491.2005.01448.x. PMID 15787679
- [Background] Phung OJ, Scholle JM, Talwar M, Coleman CI. Effect of noninsulin antidiabetic drugs added to metformin therapy on glycemic control, weight gain, and hypoglycemia in type 2 diabetes. JAMA. 2010 Apr 14;303(14):1410-8. doi: 10.1001/jama.2010.405. PMID 20388897
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] Tzoulaki I, Molokhia M, Curcin V, Little MP, Millett CJ, Ng A, Hughes RI, Khunti K, Wilkins MR, Majeed A, Elliott P. Risk of cardiovascular disease and all cause mortality among patients with type 2 diabetes prescribed oral antidiabetes drugs: retrospective cohort study using UK general practice research database. BMJ. 2009 Dec 3;339:b4731. doi: 10.1136/bmj.b4731. PMID 19959591
- [Background] Selvin E, Bolen S, Yeh HC, Wiley C, Wilson LM, Marinopoulos SS, Feldman L, Vassy J, Wilson R, Bass EB, Brancati FL. Cardiovascular outcomes in trials of oral diabetes medications: a systematic review. Arch Intern Med. 2008 Oct 27;168(19):2070-80. doi: 10.1001/archinte.168.19.2070. PMID 18955635
- [Result] Alexander GC, Sehgal NL, Moloney RM, Stafford RS. National trends in treatment of type 2 diabetes mellitus, 1994-2007. Arch Intern Med. 2008 Oct 27;168(19):2088-94. doi: 10.1001/archinte.168.19.2088. PMID 18955637